CLINICAL TRIAL: NCT05476406
Title: The Effects of äKwä Premium Skincare System on Improving Overall Skin Health and Beauty in Adults: An Exploratory Placebo-Controlled Clinical Study
Brief Title: Clinical Study to Evaluate the Impact of aKwa Skincare System on Skin Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 4Life Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSC-017-00
Record Dates: First submitted 2022-07-12; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Sin Health; Skin Hydration; Skin Wrinkles; Skin Porphyrins; Facial Skin Red Spots; Facial Skin Red Vasculature

STUDY DESIGN:
Intervention Model Description: One Active group and one Control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- äKwä Group (Experimental): participants use äKwä products daily as instructed for 30 days
  Interventions: Other: äKwä skincare system products
- Control Group (Active Comparator): participants use a competitor products daily as instructed for 30 days
  Interventions: Other: competitor products (control)

INTERVENTIONS:
Other: äKwä skincare system products — The skincare product system tested in this study was äKwä 6-step skincare system from 4Life Research USA, LLC ( https://www.4life.com/6613461/page/äKwä). Product directions state to use the following products morning and night in sequential order: First Wave Oil-to-Foam Cleanser, Glacier Glow Four-Way Toner, Precious Pool Vitamin Essence, Ripple Refine Eye Cream, and RainBurst Moisture Cream.
  Arms: äKwä Group
Other: competitor products (control) — Participants use whatever their normal daily routine of skincare products, which are commercially available competitor products from the marketplace.
  Arms: Control Group

SUMMARY:
The purpose of the study was to evaluate the effectiveness of the äKwä 6-step skincare system by measuring skin moisture level, fine lines and wrinkles, porphyrin count, red spots, and red vasculature counts over a 30-day period.

DETAILED DESCRIPTION:
The äKwä 6-step skincare system is comprised of various skincare products intended to be applied both morning and night. Some of the notable ingredients included in the product formulas are fermented green tea water, other ferments, niacinamide, antioxidants, and a variety of natural plant extracts. The purpose of the study was to evaluate the effectiveness of the äKwä 6-step skincare system by measuring skin moisture level, fine lines and wrinkles, porphyrin count, red spots, and red vasculature counts over a 30-day period.

ELIGIBILITY:
Inclusion Criteria:

* Individuals could participate who were at least 18 years old and in good health.

Exclusion Criteria:

* had allergies or contraindications to any ingredient of products,
* had a history of any acute or chronic disease that could interfere with or increase the risk of study participation
* had any medical procedures, such as laser resurfacing, or plastic surgery to the test sites within the last 12 months (including Botox, Restylyn, or other fillers)
* chronic skin allergies (dermatitis, eczema, psoriasis)
* had been treated for skin cancer within the last 12 months or have damaged skin near the facial area (e.g., sunburn, tattoos, scars, or other disfigurations)
* pregnant or planning to become pregnant in the following 12 weeks, or lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Skin Hydration | 30 days
  measure facial skin moisture level at pre-defined spots, with SkinFit instrument
Red Spot Count | 30 days
  measure the number of facial red spots at predefined areas, with SkinFit instrument
Red Vascular Count | 30 days
  measure the number of facial red vasculature at predefined areas, with SkinFit instrument
Porphyrin Count | 30 days
  measure the number of facial porphyrin at predefined areas, with SkinFit instrument
Wrinkles | 30 days
  measure the number of wrinkles and fine lines at predefined areas, with SkinFit instrument
Pores | 30 days
  measure the number of skin pores at predefined areas, with SkinFit instrument
Texture | 30 days
  measure the number of uneven skin textures, at predefined areas, with SkinFit instrument

CONTACTS AND LOCATIONS:
Overall Officials: David Vollmer, PhD, Study Chair — 4LIFE
Locations (1):
- 4Life Research, Sandy City, Utah, United States